CLINICAL TRIAL: NCT07072923
Title: Utility of Antibiotic Impregnated Beads in Lower Extremity Osteomyelitis
Brief Title: Antibiotic Impregnated Beads in Osteomyelitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Talha Riaz, MD, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005515
Record Dates: First submitted 2025-03-07; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Osteomyelitis of the Foot; Antibiotic Impregnated Beads; Osteomyelitis of Lower Extremities
Keywords: osteomyelitis, lower extremity, foot, calcium sulfate beads
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Intervention Model Description: This is a randomized, single blinded, prospective clinical trial where the treatment group will receive IV and/or oral antibiotics plus antibiotic impregnated beads, and the control group will receive IV and/or oral antibiotics plus calcium sulfate beads without antibiotics (sham beads). Systemic antibiotics therapy and the antibiotics contained in the antibiotic impregnated beads will be best available agents determined by the surgeon and infectious disease specialist.
Who Masked: Participant
Masking Description: Randomization table will be prepared with treatment allocation specified in sealed envelopes. Participants are assigned a study number sequentially after consent is obtained. The surgeon and infectious disease specialist will develop a plan for IV and/or oral antibiotics based on culture results from the initial surgery.
  In addition, they will develop a plan for local antibiotics to be incorporated in the calcium sulfate beads. Antibiotics will actually be added only if the patient is assigned to the treatment group. The Investigator will then pull the envelope for the prospective study number and obtain the assigned treatment (antibiotic loaded beads versus sham beads). The calcium sulfate beads (with or without antibiotics will be placed during the second surgical procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV and/or oral antibiotics with local antibiotic loaded calcium sulfate beads (Experimental): These will be patient who will receive active systemic antibiotics plus calcium sulfate beads loaded with antibiotics
  Interventions: Device: Calcium sulfate beads (sham beads)
- IV and/or oral antibiotics plus calcium sulfate beads without antibiotics (sham beads) (Active Comparator): These patients will receive IV and/or oral antibiotics plus sham beads. They will receive antibiotics systemically.
  Interventions: Drug: Antibiotic loaded calcium sulfate beads

INTERVENTIONS:
Drug: Antibiotic loaded calcium sulfate beads — Calcium sulfate beads will be loaded with best available antibiotics based on surgeon/infectious disease specialist determination from the following options (vancomycin, daptomycin, cefazolin, cefepime, tobramycin, amphotericin B, micafungin, and voriconazole).
  Arms: IV and/or oral antibiotics plus calcium sulfate beads without antibiotics (sham beads)
Device: Calcium sulfate beads (sham beads) — Calcium sulfate beads will be prepared without added antibiotics and placed during the second surgery.
  Arms: IV and/or oral antibiotics with local antibiotic loaded calcium sulfate beads

SUMMARY:
Lower extremity bone infections, such as osteomyelitis, often occur after bone fractures, surgery, or when prosthetic joints or hardware become infected. Treatment usually includes antibiotics, chosen based on the infection's specifics. Options include intravenous (IV) or oral antibiotics, and sometimes local treatment with antibiotic-loaded beads placed directly at the infection site. Traditionally, these beads are made of non-absorbable materials, requiring a second surgery to remove them. However, a newer approach uses absorbable calcium sulfate beads, which can deliver higher antibiotic doses and don't need removal. This study will compare the use of IV and/or antibiotics in combination with absorbable antibiotic calcium sulfate beads with IV and/or oral antibiotics without absorbable beads, which serves as the current standard of care.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of absorbable antibiotic beads in treating lower extremity (LE) infections and compare it to the current standard care. The study has several objectives: (1) to compare treatment failure rates between patients receiving intravenous (IV) and/or oral antibiotics plus antibiotic loaded absorbable beads with IV and/or oral antibiotics plus beads without antibiotics (sham beads). The primary question to be answered is whether patients treated with oral and/or IV antibiotics in conjunction with absorbable antibiotic beads have outcome (failure rate) that is not higher than those treated with standard care alone. The study's hypothesis is that the failure rate for patients receiving IV and/or oral antibiotics combined with antibiotic beads will be non-inferior to those receiving the standard care of IV or oral antibiotics without beads. The study will primarily focus on treatment failure rates as a key endpoint to measure effectiveness and compare the two treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* patients with lower extremity osteoarticular infections with or without hardware

Exclusion Criteria:

* patients who are hemodynamically unstable or have altered mental status and cannot give consent
* patient per investigators discretion are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
End of Therapy - Clinical Failure | End of Therapy (usually 4-6 weeks)
  1. Presence of at least one clinical criterium for failure (frank pus adjacent to bone or implant or draining sinus tract), OR
  2. phenotypically indistinguishable bacteria isolated from two or more deep-tissue samples or a single closed aspirate or biopsy OR
  3. histologic criteria including presence of characteristic inflammatory infiltrate or microorganisms.

IPD SHARING:
Plan to Share IPD: Undecided